CLINICAL TRIAL: NCT06915402
Title: A Post-market, Interventional, Confirmative Clinical Investigation to Evaluate the Performance and the Safety of "LMW - CL - HA - FACE/BODY" Used as Intended for the Restoration of the Physiological Volumes of the Cheeks
Brief Title: Efficacy and Safety of "LMW - CL - HA - FACE/BODY" for the Augmentation of the Cheeks
Acronym: RF-HA-FB-2024
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rose Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RF-HA-FB-2024
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Esthetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Non-comparative (Experimental): LMW - CL -HA FACE/BODY is used as intended for the restoration of the physiological volumes of the cheeks. In this study, it is planned to include 26 areas (1 area comprises both cheeks), including a drop-out rate of 10%. "LMW - CL - HA FACE/BODY" is available in a double pack containing two 2 ml syringes and for this study the package containing two 2 ml syringes will be used.
  Interventions: Device: "LMW - CL - HA FACE/BODY

INTERVENTIONS:
Device: "LMW - CL - HA FACE/BODY — The dosage to be used for the individual case is at the discretion of the doctor. The periodicity with which to repeat the procedure depends on different factors, concerning both the physiology of the patient (skin type, individual metabolism, anatomy, age) and lifestyle; another element to consider is related to the implantation techniques adopted. After the first treatment, the result can be retouched after 15 days, repeating the treatment after 9-12 months to maintain the results obtained. Local anesthesia for facial treatments can be performed, in order to ensure the necessary comfort for the patient. The area of intervention must be cleaned with antiseptic solutions before proceeding to the implant. Do not use quaternary ammonium-based disinfectants, as they can react with the HA and form precipitates."LMW - CL - HA FACE/BODY" is to be used intracutaneously and must not be injected into the blood vessels. Further details on the injection procedure are reported in the IFU.

SUMMARY:
Midface volume loss is a typical sign of facial aging. Age-related loss of subcutaneous fullness in the malar prominence results in a less healthy facial proportion. Indeed, the primary goal in any rejuvenation procedure should be to restore the balanced distribution of facial fullness that characterizes the youthful face. Rejuvenating treatments of the cheeks have a significant effect on an overall appearance and on neighbouring periorbital area, making additional treatments unnecessary. Innovative techniques to restore volume loss in the cheeks include the use of hyaluronic acid (HA) volumizing fillers created for facial sculpting. The result of such treatments is a harmonic and natural look, because the technique respects the physiologic alterations occurring during aging. HA is a natural and unbranched polymer belonging to a group of heteropolysaccharides named glycosaminoglycans. The primary structure of HA is a linear chain containing repeating disaccharide units linked by beta 1,4-glycosidic bonds. Each disaccharide consists of N-acetyl-d-glucosamine and d-glucuronic acid connected by beta-1,3-glycosidic bonds. HA is distributed ubiquitously throughout the extracellular matrix (ECM) of the skin. HA retains water to a remarkable extent; it is responsible for the hydration and viscoelasticity of the skin. As the skin ages, the content of ECM components, such as HA, decreases and this decrease directly correlates with volume loss, reduced moisture and increased rhytid formation.

HA has excellent viscoelasticity, high moisture retention capacity, and unique hygroscopic properties. In addition to its properties, HA is well-tolerated, nonimmunogenic, biocompatible, and biodegradable. For these reasons it has been widely used in a variety of biomedical applications, including aesthetic medicine. HA-based formulations are normally injected into the dermis (as dermal fillers) to restore skin volume and minimize the appearance of wrinkles and folds. An ideal soft tissue filler should also provide an optimal balance of longevity, lifting capacity and ease of injection. In this context, "LMW - CL - HA FACE/BODY" is an injectable medical device indicated for the restoration of the physiological volumes of the face and body. The main ingredient is cross-linked HA of non-animal origin, produced by bacterial fermentation at low molecular weight (100KDa).

The aim of this post-market, interventional, confirmative clinical investigation is to evaluate the performance and the safety of "LMW - CL - HA FACE/BODY" used as intended for the restoration of the physiological volumes of the cheeks

ELIGIBILITY:
Inclusion Criteria:

1. Subject Informed consent form (ICF) signed;
2. Female and male Subjects aged 18-75 years;
3. Subjects with low moderate and moderate kind of skin sagging of the face (FVLS between 2 and 4 score) desiring augmentation of both cheeks;
4. Willingness to follow all study procedures, including attending all site visits, tests and examinations;
5. Agreeing to present at each study visit without make-up;
6. Accepting to not change their habits regarding food, physical activity, make-up use, face cosmetic and cleansing products;
7. Willingness to follow indications to not be exposed to make-up, excessive heat (sun, UV tanning sessions or laser) or intense cold after the treatment and until the complete absorption of swelling and reddening.

Exclusion Criteria:

Subjects with asymmetries in the cheeks, which in the opinion of the PI could require treatment of only one side of the face, prior to study inclusion; 2. Other - different - clinical conditions of the skin (i.e. rosacea, psoriasis, vitiligo, active eczema, severe scleroderma, severe acne and diagnosticated cancer with/without ongoing antitumor therapy); 3. Botulinum toxin injections in face areas other than forehead, lips, chin within 6 months prior to study inclusion; 4. Infectious or inflammatory processes near the area of intervention or in the face in general; 5. Presence of cutaneous disease on the tested area, as malformations and recurrent facial/labial herpes; 6. Presence of tendon, bone or muscular implants near the area of intervention; 7. Presence of hypertrophic scars near the area of treatment; 8. Presence of permanent filler, of traction wires or prostheses in the face; 9. Ongoing cutaneous allergies; 10. Known hypersensitivity to cheloids; 11. Allergy or contraindications to device components; 12. Immune system illnesses/disease; 13. Uncontrolled diabetes mellitus or uncontrolled systemic diseases (endocrine, hepatic renal, cardiac, pulmonary, neurological disorder); 14. Problems with coagulation or anti-coagulating therapies in progress; 15. Treatment with substances which act on blood fluidity (e.g. Aspirin, NSAIDs, Vitamin E) within 5 days prior to study inclusion; based on Investigator's judgment cardioaspirin might be allowed; 16. Known drug and/or alcohol abuse; 17. Mental incapacity that precludes adequate understanding or cooperation; 18. Any previous permanent and non-permanent cutaneous treatment for aesthetic correction (biomaterial implant, lifting, laser, chemical peeling, fillers) of the face within 6 months prior to study inclusion; 19. Pregnancy or breastfeeding; 20. Dental pathologies: tooth decay, abscesses, preparation for implants; 21. Participation in another investigational study within 1 month prior to study inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the performance of the filler LMW - CL - HA FACE/BODY used as intended for the restoration of the physiological volumes of the cheeks after 6 months compared to baseline volume. Change will be assessed. | V0 (Screening/Base line (V0) and V3 (End of Study) 6 months from V0
  To evaluate the performance of the filler LMW - CL - HA FACE/BODY used as intended for the restoration of the physiological volumes of the cheeks in patients requiring cheeks augmentation. The change from baseline will be assessed by the physician and Facial Volume Loss Scale (FVLS) will be used at the end of the study (V3). For evaluation of FVLS photographs will be taken using a 2D camera according to standardized and reproducible procedures. The FVLS includes five gradations. The face is assessed according to three criteria: contour, bony prominence, and visibility of musculature. Scale grades are:
  Grade 1. Mild flattening or shadowing of one or more facial regions; Grade 2: An intermediate point between Grade 1 and Grade 3. Grade 3: Moderate concavity of one or more facial regions. Grade 4: An intermediate point between Grade 3 and Grade 5. Grade 5: Severe indentation of one or more facial regions.

SECONDARY OUTCOMES:
To evaluate the performance of the filler LMW - CL - HA FACE/BODY used as intended for the restoration of the physiological volumes of the cheeks during all the study visits by Facial Volume Loss Scale | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0) V2 (3 months from V0) V3 (6 months from V0).
  The FVLS includes five gradations. The face is assessed according to three criteria: contour, bony prominence, and visibility of musculature. Scale grades are: Grade 1. Mild flattening or shadowing of one or more facial regions (including the cheek, temple, preauricular, and periorbital areas); no prominent bony landmarks; no visibility of underlying musculature. Grade 2: An intermediate point between Grade 1 and Grade 3. Grade 3: Moderate concavity of one or more facial regions (including the cheek, temple, preauricular, and periorbital areas); prominence of bony landmarks; may have visibility of underlying musculature. Grade 4: An intermediate point between Grade 3 and Grade 5. Grade 5: Severe indentation of one or more facial regions (including the cheek, temple, preauricular, and periorbital areas); severe prominence of bony landmarks; clear visibility of underlying musculature.
To evaluate the performance of the filler LMW - CL - HA FACE/BODY to improve aesthetic appearance by GAIS at baseline and follow-up visits | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0) V2 (3 months from V0) V3 (6 months from V0)
  the Global Aesthetic Improvement Scale (GAIS) scale will be assessed. The GAIS will be completed independently by both the Subject and the physician. The GAIS is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator. The rating categories were "worse," "no change," "improved," "much improved," and "very much improved."
To evaluate pain intensity after injection of LMW - CL - HA FACE/BODY | V0 (Baseline visit day 0, IP administration)
  A Numerical Rating Scale (NRS) will be administered to the Subject at V0. The numeric rating scale is a scale designed to help assess the extent of an individual's pain and improve communication regarding pain with health care providers. This scale can help guide the diagnostic process, track the progression of the pain, and more. Numeric pain rating scale, which measures 0-10 - with 0 as no pain and 10 as the worst pain imaginable.
To evaluate Subject satisfaction after 6 months from baseline. | V3 (6 months from V0)
  To evaluate Subject satisfaction after 6 months from baseline, a 5 Likert Scale will be completed by the Subject at EOS visit (V3). The Likert scale is a five point scale that is used to allow an individual to express how much they agree or disagree with a particular statement. Here's a breakdown of a typical 5-point Likert scale:
  1. Strongly Disagree
  2. Disagree
  3. Neutral (or Neither Agree nor Disagree)
  4. Agree
  5. Strongly Agree This scale allows respondents to express the intensity of their feelings towards a given statement, making it easier to quantify subjective data. It's widely used because it's simple to understand and analyze.
To evaluate the safety and tolerability of LMW - CL - HA FACE/BODY | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0) V2 (3 months from V0) V3 (6 months from V0)
  Facial examination (e.g., reddening, oedema, itching and pain in the touch, bruising, hardening or nodules at the injection site, coloring and discoloring of the skin at the point of injection) will be assessed at each visit

OTHER OUTCOMES:
Assessment of Device Deficiency/Incidents. | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0)
  Device deficiency/incident information will be collected by the investigator or its delegates on the CRF's.
Safety will be monitored through the reporting of the adverse events, serious adverse events and concomitant medications during the entire study duration. | V0 (Baseline visit day 0, IP administration) V1 (15 days from V0) V2 (3 months from V0) V3 (6 months from V0)
  The event, date of onset, severity, duration, and relationship to the device will be recorded. Subjects will receive a diary to record any deviation from the normal health status as well as any concomitant medication taken.

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Parodi, Dr. med., Principal Investigator — Ospedale Regionale di Lugano- Servizio di Chirurgia Plastica, Ricostruttiva ed Estetica EOC Ospedale Regionale di Lugano Via Pietro Capelli 1 CH-6962 Vi-ganello